CLINICAL TRIAL: NCT03282539
Title: Lumen Apposing Metal Stents With and Without a Coaxial Double Pigtail Stent in the Management of Pancreatic Fluid Collections
Brief Title: Lumen Apposing Metal Stents With and Without a Double Pigtail Stent in Pancreatic Collections
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, JOAN B GORNALS, PhD, Hospital Universitari de Bellvitge
Other Study IDs: LAMSpig1
Record Dates: First submitted 2017-08-08; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Collection
Keywords: Lumen apposing metal stents; Double pigtail stents; Endoscopic ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- LAMS: EUS-guided transmural drainage of pancreatic fluid collections with lumen apposing metal stents.
  Interventions: Device: LAMS
- LAMS + pigtail: EUS-guided transmural drainage of pancreatic fluid collections with lumen apposing metal stents and a coaxial double pigtail stent
  Interventions: Device: LAMS + pigtail

INTERVENTIONS:
Device: LAMS — EUS-guided transmural drainage of pancreatic fluid collections with lumen apposing metal stents
  Groups: LAMS
Device: LAMS + pigtail — EUS-guided transmural drainage of pancreatic fluid collections with lumen apposing metal stents and a coaxial double pigtail stent
  Groups: LAMS + pigtail

SUMMARY:
The study evaluates the security of LAMS with ando without a coaxial double pigtail plastic stent in the management of pancreatic fuid collections.

DETAILED DESCRIPTION:
The introduction of lumen-apposing metal stents (LAMS) represented a great improvement in the EUS-guided transmural drainage of pancreatic fluid collections (PFCs). It is postulated safer than other types of stents due to the presence of bilateral anchoring flanges, designed to appose the stomach or duodenum to the PFC wall minimizing the risk of perforation or peritoneal leakage. In addition, the larger lumen diameter facilitates the drainage of PFC, specially the walled-off pancreatic necrosis (WOPN). However, secondary adverse effects such as infection due to complete or partial stent obstruction, migration, bleeding or buried LAMS syndrome have also been related . The placement of a coaxial double pigtail plastic within the LAMS has been reported beneficial in order to avoid external migration or the lumen obstruction and to the prevention of bleeding and other adverse events. The aim of this study was to evaluate the efficacy and safety of LAMS with and without a coaxial double pigtail plastic stent in the EUS-guided transmural drainage of PFCs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic fluid collections and indication of drainage.
* EUS-guided trasmural drainage wiht lumen apposing metal stents.
* Criteria for drainage were as specified by the Working Group of the International Association of Pancreatology.

Exclusion Criteria:

* Other types of collections and stents
* Severe coagulopathy (protombin time > 1,5) or thrombocytopenia (platelet count < 50 x 109/L)
* PFCs with a previous attempt failed of EUS-guided transmural drainage
* Age younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients wiht pancreatic fluid collections and indication for EUS-guided transmural drainage in accordance l wiht international creteria.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | Outcomes will be assessed 6 months after the inclusion of last patient.
  Defined and graded according to the ASGE lexicon's severity grading system

CONTACTS AND LOCATIONS:
Overall Officials: Joan Gornals, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
The results of the stuydy will be shared with other researchers.